CLINICAL TRIAL: NCT01757847
Title: Acceptance-based Group Intervention for Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F7400-R
Record Dates: First submitted 2012-12-11; First posted 2012-12-31 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-10

CONDITIONS: Binge-Eating Disorder
Keywords: Binge-Eating Disorder; Obesity; emotional eating
MeSH Terms: conditions — Binge-Eating Disorder; Obesity; Emotional Eating | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief MOVE-II active control group intervention (Active Comparator): The MOVE-II protocol was designed to reinforce the weight-loss principles that patients learn in MOVE! and to provide support in continued weight loss. This protocol includes a psycho-educational component that reinforces the key information from the medical, nutrition, and weight loss strategies modules of the MOVE! program. After review of the psycho-educational components, patients have the opportunity to share their challenges with binge eating and weight loss. Patients will then be able to receive support and feedback from other group members and the therapist. In addition, the active control group focuses on increasing self-esteem and self-efficacy by exploring patient strengths and maintaining therapeutic alliance and optimism. The brief MOVE-II active control group protocol will be delivered in four 2-hour weekly group sessions to patient with overweight or obesity who have completed the VA San Diego MOVE program.
  Interventions: Behavioral: Brief MOVE-II control group intervention
- Acceptance and Commitment Therapy (ACT) (Experimental): Acceptance and Commitment Therapy (ACT), has been effective in reducing distress, increasing quality of life, and improving other indices of health in a wide range of conditions from depression to diabetes. The ACT protocol for this study focuses on reducing binge eating and distress and improving functioning in individual who are overweight or obese. The protocol focuses on a) thoughts, feelings, and bodily sensations in the context of efforts to lose weight; b) limitations of efforts to control or eliminate negative thoughts or emotions, stress, or food cravings; c) changing expectations and goals from elimination of stress or cravings to living as well as possible with such feelings; d) mindfulness exercises to increase awareness; and e) identification of personal values and goals to achieve improved quality of life. The protocol will be delivered in four 2-hour weekly group sessions to patients with overweight or obesity who have completed the VA San Diego MOVE program.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — The ACT group protocol consists of four 2-hour weekly sessions focusing on a) thoughts, feelings, and bodily sensations in the context of efforts to lose weight; b) limitations of efforts to control or eliminate negative thoughts or emotions, stress, or food cravings; c) changing expectations and goals from elimination of stress or cravings to living as well as possible with such feelings; d) mindfulness exercises to increase awareness; and e) identification of personal values and goals to achieve improved quality of life.
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy (ACT)
Behavioral: Brief MOVE-II control group intervention — The MOVE-II protocol was designed to reinforce the weight-loss principles that patients learn in MOVE! and to provide support in continued weight loss. The brief MOVE-II active control group protocol will be delivered in four 2-hour weekly group sessions. This protocol includes a psycho-educational component that reinforces the key information from the medical, nutrition, and weight loss strategies modules of the MOVE! program. After review of the psycho-educational components, patients have the opportunity to share their challenges with binge eating and weight loss. Patients will then be able to receive support and feedback from other group members and the therapist. In addition to reinforcing the strategies taught during MOVE! and to provide support in implementing those strategies, the active control group focuses on increasing self-esteem and self-efficacy by exploring patient strengths and maintaining therapeutic alliance and optimism.
  Arms: Brief MOVE-II active control group intervention

SUMMARY:
This study proposes to compare a brief Acceptance and Commitment Therapy (ACT) group intervention to an active control group in a sample of 154 overweight or obese binge eating Veterans who have completed the VA's national behavioral weight management program (MOVE!). This study anticipates that the ACT intervention will reduce binge eating and distress while improving functioning and maintenance of weight loss.

DETAILED DESCRIPTION:
Approximately two-thirds of all adults and close to 75% of Veterans are overweight or obese, making obesity a national epidemic with significant impairments in physical and psychological functioning, increasing healthcare costs, and high mortality rates. A significant proportion of overweight and obese individuals binge eat in response to stress or negative emotions, further contributing to obesity. Obesity and binge eating are independently related to a number of physical and mental health co-morbidities such as diabetes, coronary heart disease, osteoarthritis, respiratory symptoms, depression, and anxiety. Although behavioral weight loss interventions have been partially effective, few show long-term maintenance of weight loss, especially for patients with binge eating behavior. Thus, a stepped-care approach that provides more intensive treatment to specifically address the emotional and behavioral factors associated with problematic eating and obesity may be necessary. Acceptance and Commitment Therapy (ACT), an empirically-supported intervention that is being rolled out nationally by the VA, has been effective in reducing distress, increasing quality of life, and improving other indices of health in a wide range of conditions from depression to diabetes. The investigator's preliminary findings suggest that a brief ACT-based group intervention for patients with overweight or obesity can substantially reduce binge eating and distress, and improve functioning. This study proposes to test the efficacy of an ACT intervention for binge eating in conjunction with a standard behavioral weight loss intervention, Managing Overweight and/or Obesity for Veterans Everywhere (MOVE!), at the VA San Diego Healthcare System (VASDHS). Patients (N = 154) who are overweight or obese (body mass index > 25 kg/m2) and meet the clinical criteria for binge eating will be randomized to receive either four 2-hour weekly ACT intervention groups or brief MOVE-II active control groups after their participation in MOVE!. This study hypothesizes that: 1) patients in the ACT intervention will experience significantly greater reductions in binge eating severity than patients in the brief MOVE-II active control group (primary outcome); 2) patients in the ACT intervention will experience significantly greater improvements in physical and mental health functioning, obesity-related quality of life, physical activity levels, caloric and nutrient intake, emotional distress symptoms, binge frequency, and other forms of emotional eating than patients in the brief MOVE-II active control group; 3) gains associated with the ACT intervention will be maintained longer than gains associated with the brief MOVE-II active control group; 4) at 3-month and 6-month follow-ups, patients in the ACT intervention will have greater decreases in body mass index compared to patients in the brief MOVE-II active control group; and 5) measures of acceptance and action will mediate treatment response in the ACT intervention on outcomes of interest. Given the significant physical and psychological sequelae of binge eating and obesity, a brief intervention that can reduce disordered eating, enhance the maintenance of weight loss, and improve functioning among patients who suffer from binge eating, could be critical in the comprehensive approach to patient care at the VA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overweight or obesity (i.e., BMI > 25 kg/m2), as verified by a study physician after a medical evaluation and examination of medical records;
* Attendance of at least 60% of weight loss sessions of the MOVE! program (i.e., 5 of 8 sessions).
* At least 18 years old

Exclusion Criteria:

* Serious or unstable medical or psychiatric illness (i.e., current unmanaged psychosis, manic episode, anorexia nervosa, bulimia nervosa, or substance abuse within the past year) or psychosocial instability (e.g., homelessness) that could compromise study participation;
* Conditions in which exercise or weight loss will be detrimental to one's health (e.g., pregnancy);
* Active suicidal ideation or history of suicide attempt within 5 years;
* Pharmacotherapy for obesity (e.g., Orlistat or Meridia) or bariatric surgery within the past 6 months or planning to start such treatments in the next 6 months;
* Current participation in group or individual psychotherapy for weight management or binge eating;
* Previous treatment with ACT;
* Unwillingness to agree not to change professionally delivered mood treatments and psychotherapy (e.g., begin new therapy or group; discontinue a treatment; increase the dose of medication) for the duration of 4-week study treatment period unless medically necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niloofar Afari, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not available for data sharing but aggregate data may be available by contacting the PI.

REFERENCES:
- [Derived] Morse JL, Fishbein JN, Wooldridge JS, Herbert MS, Afari N. Posttraumatic Stress Disorder and Weight Loss in Male and Female Active-duty Service Members: A Weight Management Study. Mil Med. 2025 Sep 1;190(9-10):e1784-e1791. doi: 10.1093/milmed/usae561. PMID 39797515
- [Derived] Afari N, Herbert MS, Godfrey KM, Cuneo JG, Salamat JS, Mostoufi S, Gasperi M, Ober K, Backhaus A, Rutledge T, Wetherell JL. Acceptance and commitment therapy as an adjunct to the MOVE! programme: a randomized controlled trial. Obes Sci Pract. 2019 Aug 16;5(5):397-407. doi: 10.1002/osp4.356. eCollection 2019 Oct. PMID 31687165

RESULTS

PARTICIPANT FLOW:
Groups:
- Brief MOVE-II Active Control Group Intervention: The MOVE-II protocol was designed to reinforce the weight-loss principles that patients learn in MOVE! and to provide support in continued weight loss. The brief MOVE-II active control group protocol was delivered in four 2-hour weekly group sessions. This protocol includes a psycho-educational component that reinforces the key information from the medical, nutrition, and weight loss strategies modules of the MOVE! program. After review of the psycho-educational components, patients have the opportunity to share their challenges with binge eating and weight loss. Patients will then be able to receive support and feedback from other group members and the therapist. In addition, the active control group focuses on increasing self-esteem and self-efficacy.
Period: Overall Study
Arm/Group | Brief MOVE-II Active Control Group Intervention | Acceptance and Commitment Therapy (ACT)
Started | 44 | 46
Completed | 41 | 42
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief MOVE-II Active Control Group Intervention | Acceptance and Commitment Therapy (ACT) | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.52 (9.33) | 56.23 (10.34) | 56.87 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 37 | 33 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 42 | 40 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 7 | 17
  White | 32 | 36 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 44 | 46 | 90
Binge Eating Scale [Mean (Standard Deviation); unit: units on a scale] — This measure contains 16 questions that describe both behavioral and emotional manifestations of a binge episode. This scale was specifically developed to assess binge eating severity and associated emotional distress in overweight and obese individuals. The total score for the measure ranges from 0-46 points with higher scores indicating greater problems with binge eating and lower scores indicating better outcome.
  units on a scale | 17.48 (8.25) | 15.53 (9.28) | 16.47 (8.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Binge Eating Scale (BES) at 4 Weeks, 3 Months and 6 Months
Description: This measure contains 16 questions that describe both behavioral and emotional manifestations of a binge episode. This scale was specifically developed to assess binge eating severity and associated emotional distress in overweight and obese individuals. The total score for the measure ranges from 0-46 points with higher scores indicating greater problems with binge eating and lower scores indicating better outcome.
Time Frame: post treatment (4 weeks), 3 months, 6 months
Population: participants with measurement at baseline and at least one other time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief MOVE-II Active Control Group Intervention | Acceptance and Commitment Therapy (ACT)
Number analyzed (Participants) | 42 | 43
units on a scale
  Baseline | 17.38 (8.15) | 15.45 (9.19)
  Post treatment | 10.52 (7.29) | 13.52 (9.05)
  3 month follow up | 10.47 (7.40) | 11.90 (8.65)
  6 month follow up | 10.00 (7.49) | 12.20 (7.32)

2. Secondary Outcome: Change From Baseline in The Obesity-related Well Being Scale (ORWELL-97) at 4 Weeks, 3 Months, and 6 Months
Description: The ORWELL-97 is a self-report measure of obesity-related quality of life. It has been validated on obese patients. The total score ranges from 0-162 with higher scores indicating lower quality of life and decreasing scores indicating improvement in the outcome.
Time Frame: post treatment (4 weeks), 3 months, 6 months
Population: Participants with measurement at baseline and at least one other time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief MOVE-II Active Control Group Intervention | Acceptance and Commitment Therapy (ACT)
Number analyzed (Participants) | 42 | 43
units on a scale
  Baseline | 50.17 (28.26) | 49.47 (30.60)
  Post Treatment | 41.86 (22.65) | 46.02 (33.57)
  3 month follow up | 41.07 (26.77) | 38.79 (29.14)
  6 month follow up | 37.90 (31.87) | 36.55 (27.82)

ADVERSE EVENTS:
Time Frame: Duration of study up to the 6-month follow-up.
Arm/Group | Brief MOVE-II Active Control Group Intervention | Acceptance and Commitment Therapy (ACT)
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 0/44 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No